CLINICAL TRIAL: NCT00865969
Title: A Multicenter, Open-Label Trial of Belinostat in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: Belinostat in Relapsed or Refractory Peripheral T-Cell Lymphoma
Acronym: PTCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-19; 2008-005843-40 (EudraCT Number)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Belinostat; Peripheral T-cell lymphoma; PXD101; PTCL; HDAC inhibitor; Histone deacetylase inhibitor
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — belinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belinostat (Experimental): Belinostat 1000 mg/m^2 administered as a 30 minute IV infusion on Days 1-5 of every 3-week cycle until disease progression or unmanageable treatment-related toxicities.
  Interventions: Drug: Belinostat

INTERVENTIONS:
Drug: Belinostat
  Other Names: PXD101

SUMMARY:
The purpose of this study is to assess efficacy and safety of belinostat in participants with relapsed or refractory peripheral T-cell lymphoma (PTCL), who failed at least one prior systemic therapy.

DETAILED DESCRIPTION:
This is an open-label, multicenter, single arm efficacy and safety study in participants with relapsed or refractory peripheral T-cell lymphoma, who have failed at least one prior systemic therapy.

Approximately 120 participants will be enrolled. Participants will be treated with 1000 mg/m^2 belinostat administered as a 30-minute IV infusion on Days 1-5 of every 3-week cycle until there is disease progression or unmanageable treatment-related toxicities.

The primary study endpoint is objective response rate (ORR) based on the International Harmonization Project (IHP) revision International Working Group (IWG) criteria. Safety will be evaluated during the study and for 30 days after the last administration of study drug. Adverse events and laboratory studies will be graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v. 3.0.

ELIGIBILITY:
Inclusion criteria:

* A histologically confirmed diagnosis of PTCL
* Participants must have relapsed or refractory disease after at least one prior systemic anticancer regimen. Systemic anticancer therapy is defined as chemotherapy or immunotherapy administered systemically.
* Participants must have at least one site of disease measurable in two dimensions by computed tomography (CT).
* Age ≥ 18 years.
* Adequate bone marrow, liver, and renal functions.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Negative pregnancy test for women of childbearing potential.

Exclusion criteria:

* Relapse within 100 days of autologous or allogeneic bone marrow transplant.
* Prior histone deacetylase (HDAC) inhibitor therapy.
* Co-existing active infection or any medical condition likely to interfere with trial procedures.
* Severe cardiovascular disease.
* Clinically significant central nervous system disorders with altered mental status or psychiatric disorders precluding understanding of the informed consent process and/or completion of the necessary studies.
* Active concurrent malignancy (except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix).
* Symptomatic or untreated central nervous system (CNS) metastases.
* Pregnant or breast-feeding women.
* Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2013-11-05 (Actual); Study Completion 2014-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Brown, MD, Principal Investigator — H:S Rigshospitalet, Department of Hematology, Denmark; Pier L Zinzani, MD, Principal Investigator — Università di Bologna, Italy; André Bosly, MD, Principal Investigator — Cliniques Universitaires UCL Mont Godinne, Belgium; Georges Fillet, MD, Principal Investigator — University of Liege, Belgium; Eric van den Neste, MD, Principal Investigator — Clinique Universitaier Saint Luc, Belgium; Nicolas Monier, MD, Principal Investigator — Hôpital de l'Archet 1 Centre Hospitalier Universitaire (CHU) de Nice, France; Elisabeth Perez, MD, Principal Investigator — Groupe Hospitalier Sud Réunion, France; Maria Delioukina, MD, Principal Investigator — City of Hope National Medical Center, USA; Adam Lerner, MD, Principal Investigator — Boston Medical Center, USA; Lydia Dreosti, MD, Principal Investigator — Pretoria Academic Hospital, South Africa; D. Moodley, MD, Principal Investigator — Drs Pirjol, Szpak and Moodley Inc, Durban, South Africa; Hanneke C. Kluin-Nelemans, MD, Principal Investigator — University Medical Center Groningen UMCG, The Netherlands; G. Sissolak, MD, Principal Investigator — Tygerberg Hospital, Cape Town, South Africa; L. Verdonk, MD, Principal Investigator — Isala Clinics, Zwolle, The Netherlands; O. Visser, MD, Principal Investigator — VU Medical Center, Amsterdam, The Netherlands; Owen A. O'Connor, MD, Principal Investigator — New York University Cancer Institute, USA; Sarit Assouline, MD, Principal Investigator — McGill University, Department of Oncology Clinical Research Program, Montreal, Canada; Juan Manuel Sancho Cia, MD, Principal Investigator — ICO Hospital Germans Trias i Pujol, Badalona, Spain; Consolación Rayon, MD, Principal Investigator — Hospital Universitario Central de Asturias, Oviedo, Spain; Sonia Gonzales, MD, Principal Investigator — Hospital Clinico Universitario de Santiago, Santiago de Compostella, Spain; Lorenz Trümper, MD, Principal Investigator — Universität Göttingen, Abteilung Hämatologie und Onkologie, Göttingen, Germany; Andreas Viardot, MD, Principal Investigator — Universitätsklinikum Ulm, Ulm, Germany; Georg Hess, MD, Principal Investigator — Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Germany; Hans-Heinrich Wolf, MD, Principal Investigator — Universitätsklinikum (AöR) der Martin-Luther-Universität Halle-Wittenberg, Halle, Germany; Andreas Neubauer, MD, Principal Investigator — University Hospital Marburg, Marburg, Germany; Michele Frank, MD, Principal Investigator — Cascade Cancer Center; Madeleine Duvic, MD, Principal Investigator — UT - M. D. Anderson Cancer Center; Andrei Shustov, MD, Principal Investigator — Fred Hutchinson Cancer Research Center - Seattle Cancer Care Alliance; Melissa Runge-Morris, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Nalini Janakiraman, MD, Principal Investigator — Henry Ford Health System; Amanda Cashen, MD, Principal Investigator — Wasington University School of Medicine- Division of Oncology; Beata Holkova, MD, Principal Investigator — Massey Cancer Center; Mohammad Tirgan, MD, Principal Investigator — Hematology Associates; Bernard Poiesz, MD, Principal Investigator — Upstate Medical Univeristy Syracuse; Charles Farber, MD, Principal Investigator — Morristown Memorial Hospital; Zale Bernstein, MD, Principal Investigator — Erie County Medical Center (Roswell Park); Ralph Boccia, MD, Principal Investigator — Center for Cancers and Blood Disorders; David Grinblatt, MD, Principal Investigator — Kellogg Cancer Care Center; Laura Blakely, MD, Principal Investigator — Accelerated Community Oncology Reseaerch Network, Inc. (ACORN); David Dennis, MD, Principal Investigator — Boca Raton Clinical Research Associates; Fernando Camacho, MD, Principal Investigator — Bronx River Medical Associates, PC; Eliot Epner, MD, Principal Investigator — Penn State Hershey Cancer Institute
Locations (117):
- United States (42):
  - City of Hope National Medical Center, Duarte, California
  - Wilshire Oncology Medical Group, Inc, La Verne, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Yale Cancer Center-Section of Medical Oncology, New Haven, Connecticut
  - Oncology Associates of Bridgeport, Trumbull, Connecticut
  - Boca Raton Clinical Research Associates, Boca Raton, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Kellogg Cancer Care Center, Evanston, Illinois
  - Illinois Cancer Specialists/Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Center for Cancers and Blood Disorders, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Northern New Jersey Cancer Associates, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Erie County Medical Center (Roswell Park), Buffalo, New York
  - Monter Cancer Center, Lake Success, New York
  - New York University Cancer Institute, New York, New York
  - New York University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Upstate Medical Univeristy Syracuse, Syracuse, New York
  - Bronx River Medical Associates, PC, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hematology Associates, Bedford, Ohio
  - St Luke's Cancer Center, Bethlehem, Pennsylvania
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Center, Sioux Falls, South Dakota
  - Associates In Oncology and Hematology, Chattanooga, Tennessee
  - University of Tennessee Cancer Institute, Knoxville, Tennessee
  - Accelerated Community Oncology Reseaerch Network, Inc. (ACORN), Memphis, Tennessee
  - UT - M. D. Anderson Cancer Center, Houston, Texas
  - The UT Health Science Centre at San Antonio, San Antonio, Texas
  - Massey Cancer Center, Richmond, Virginia
  - Cascade Cancer Center, Kirkland, Washington
  - Fred Hutchinson Cancer Research Center - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (7):
  - ZNA Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
  - AZ St. Jan, Bruges
  - Clinique Universitaire Saint Luc, Service Hématologie, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - University of Liege, Divisions of Hematology and Medical Oncology, Liège
  - Cliniques Universitaires UCL Mont Godinne, Service Hématologie, Yvoir
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - CHA Hôpital de l'Enfant-Jésus, Québec, Quebec
  - McGill University, Montreal
- Croatia (4):
  - CHC Split Clinic of Internal Diseases, Split
  - CHC Zagreb Clinic of Internal Diseases, Zagreb
  - UH Dubrava Clinic of Internal Diseases, Zagreb
  - CHC Rijeka, Clinic of Internal Diseases, Zagreb
- H:S Rigshospitalet, The Finsen Centre, KAT, Haematology Department 4241, Copenhagen, Denmark
- France (2):
  - Hôpital de l'Archet, Centre Hospitalier Universitaire (CHU) de Nice, Hématologie Clinique, Nice
  - Groupe Hospitalier Sud Réunion, Site Saint-Pierre, Saint-Pierre
- Germany (13):
  - Klinik Essen Süd, Evangelisches Krankenhaus, Essen
  - Leitender Oberarzt/Klinik für Onkologie und Hämatologie, Frankfurt
  - Universität Göttingen, Abteilung Hämatologie und Onkologie, Göttingen
  - Universitätsklinikum (AöR) der Martin-Luther-Universität Halle-Wittenberg, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätsmedizin der johannes Gutenberg -Universität Mainz, Mainz
  - University Hospital Marburg, Marburg
  - Münchner Studienzentrum Klinikum Rechts der Isar, München
  - Klinikum Nuernberg Nord, Nuremberg
  - Universitätsklinikum Rostock, Rostock
  - Universitätsklinikum Ulm, Ulm
- Hungary (4):
  - Szt István és Szt. Laszlo, Budapest
  - Belgyógyászati Klinika, Debrecen
  - Belgyógyászati Klinika Györ, Győr
  - Belgyógyászati Klinika es Kardiologial Központ, Szeged
- Israel (4):
  - The Soroka University Medical Center, Beersheba
  - Rambam Medical Center Department of Hematology, Haifa
  - Hadassah University Hospital Sharet Building Department of Hematology, Jerusalem
  - Rabin Medical Center Belinson Campus, Petah Tikva
- Italy (2):
  - Ospedale Sant'Orsola, Instituto di Ematologia e Oncologia Medica, Bologna
  - Ospedale Policlinico Careggi, Florence
- Netherlands (4):
  - VU Medical Center, Department of Haematology, Amsterdam
  - University Medical Center Groningen UMCG, Department of Haematologie, Groningen
  - Erasmus University Medical Center, Rotterdam
  - Isala Clinics, Department of Haematololgy, Zwolle
- Poland (8):
  - Klinika Nowotworów Ukladu Chlonnego Centrum Onkologii Instytut Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne Klinika Hematologii i Transplantologii, Gdansk
  - Małopolskie Centrum Medyczne, Krakow
  - Wojewódzki Szpital Specjalistyczny im M. Kopernika w Łodzi Oddział Hematologii - Klinika Hematologii, Lodz
  - Szpital Wojewódzki w Opolu/Oddział Hematologii, Opole
  - MTZ Clinical Research Sp z o.o., Warsaw
  - Instytut Hematologii i Transfuzjologii Klinika Hematologii, Warsaw
  - Wojskowy Instytut Medyczny Klinika Chorób/Wewnętrznych i Hematologii Centralnego Szpitala, Warsaw
- Russia (3):
  - State Therapeutical and Prophylactic Institution Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Russian Cancer Research Centre named after N.N. Blokhin of Russian Academy of Medical Sciences, Moscow
  - Research Center of Haematology, Moscow
- Slovakia (2):
  - Narodny Onkologicky Ustav (NOU), Bratislava
  - Klinika Hematologie a Onkohematologie FNLP a LF UPJS, Košice
- South Africa (4):
  - Tygerberg Hospital, Department of Radiation Oncology, Bellville
  - Drs pirjol, Szpak and Moodley Inc., Durban
  - Medical Oncology 2nd Floor Radiotherapy building Steve Biko Academic Hospital, Pretoria
  - Pretoria Academic Hospital, Department of Radiation Oncology, Pretoria
- Spain (8):
  - Complexo Hospitalario a Coruna, A Coruña
  - Hospital Clinico Universitario de Santiago, A Coruña
  - ICO Hospital Germans Trias i Pujol, Badalona
  - Hospital Duran i Reinals, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital General Universitario Gregorio Maranón, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
- United Kingdom (6):
  - St James's Institute of Oncology Bexley Wing, Leeds
  - Leicester Royal Infirmary, Leicester
  - Institute of Cancer/ Centre for Medical Oncology/Barts and The London School of Medicine and Dentistry, London
  - The Christie NHS Foundation Trust, The Christie Hospital,, Manchester
  - Northern Centre for Cancer Care, Freeman Hospital, Newcastle upon Tyne
  - The Royal Marsden Haemato-Oncology Wards, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campbell P, Thomas CM. Belinostat for the treatment of relapsed or refractory peripheral T-cell lymphoma. J Oncol Pharm Pract. 2017 Mar;23(2):143-147. doi: 10.1177/1078155216634178. Epub 2016 Jun 23. PMID 26921086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with relapsed or refractory T-Cell lymphoma who signed the informed consent form and met all Inclusion/Exclusion criteria were enrolled in the study.
Groups:
- Belinostat: Belinostat 1000mg/m^2 administered as a 30 minute IV infusion from Days 1-5 of a 3-week cycle until disease progression or unmanageable treatment-related toxicities.
Period: Overall Study
Arm/Group | Belinostat
Started | 129
Completed | 129
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who were received at least 1 dose of belinostat.
Arm/Group | Belinostat
Number analyzed (Participants) | 129
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with a complete response (CR) or a partial response (PR) according to International Working Group (IWG) criteria. The response was assessed based on clinical and radiological criteria. CR is defined as the disappearance of all evidence of disease. PR is defined as a regression of measurable disease and no new sites. As pre-defined, the primary endpoint analysis for this study was based on the Independent Review Committee (IRC) assessment of response.
Time Frame: 24 months
Population: Efficacy Analysis Dataset included participants who received at least 1 dose of belinostat and had a confirmed peripheral T-cell lymphoma (PTCL) diagnosis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Belinostat
Number analyzed (Participants) | 120
percentage of participants | 25.8 [18.3 to 34.6]

2. Secondary Outcome: Time to Response
Description: Time to response was defined as the time (in weeks) from first administration of treatment until first response. Response is defined as complete response (CR) or partial response (PR). CR is defined as the disappearance of all evidence of disease. PR is defined as a regression of measurable disease and no new sites.
Time Frame: 24 months
Population: Efficacy Analysis Dataset included participants who received at least 1 dose of belinostat and had a confirmed PTCL diagnosis. Overall number of participants analyzed included responding participants (CR/PR) only.
Measure: Median (Full Range); unit: weeks
Arm/Group | Belinostat
Number analyzed (Participants) | 31
weeks | 5.6 [4.3 to 50.4]

3. Secondary Outcome: Duration of Response
Description: The Duration of Response was assessed by IWG criteria per the IRC from the date the measurement criteria were first met for CR or PR (whichever status was recorded first) until the first subsequent date that relapse or progression was documented. It was estimated by the Kaplan-Meier method. Response is defined as complete response (CR) or partial response (PR). CR is defined as the disappearance of all evidence of disease. PR is defined as a regression of measurable disease and no new sites.
Time Frame: 24 months
Population: Efficacy Analysis Dataset included participants who received at least 1 dose of belinostat and had a confirmed PTCL diagnosis. Overall number of participants analysed included responding participants (CR/PR) only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belinostat
Number analyzed (Participants) | 31
months | 13.6 [4.5 to 29.4]

4. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time (in months) from first administration of treatment to the date of disease progression based on tumor assessments made according to the IWG criteria as assessed by the IRC. The progression is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: 24 months
Population: Efficacy Analysis Dataset included participants who received at least 1 dose of belinostat and had a confirmed PTCL diagnosis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belinostat
Number analyzed (Participants) | 120
months | 2 [1.5 to 2.9]

5. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) was the duration of time from first administration of study treatment to date of first documented progression or death from any cause. It was based on tumor assessments made according to the IWG criteria as assessed by the IRC. The progression is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: 24 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belinostat
Number analyzed (Participants) | 120
months | 1.6 [1.4 to 2.7]

6. Secondary Outcome: Overall Survival
Description: Overall Survival was the time from first administration of study treatment until the date of death.
Time Frame: 24 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belinostat
Number analyzed (Participants) | 120
months | 7.9 [6.1 to 13.9]

7. Secondary Outcome: Number of Participants With At Least One Serious Treatment-Emergent Adverse Event (TEAE)
Description: A TEAE was defined as an event with an onset date and time on or after the first dosing start date and time, or on or after the first dosing start date if the onset time was missing. A serious TEAE was any untoward medical occurrence that at any dose results in death, prolonged hospitalization, persistent or significant disability or congenital abnormalities.
Time Frame: 24 months
Population: Full Analysis Dataset included all participants who received at least 1 dose of belinostat.
Measure: Count of Participants; unit: Participants
Arm/Group | Belinostat
Number analyzed (Participants) | 129
Participants | 61

8. Other Pre Specified Outcome: Population Pharmacokinetics
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 25 months
Description: Participants were carefully monitored for all adverse events that occurred from the time Informed Consent was obtained until 30 days after the last study drug administration.
Arm/Group | Belinostat
All-Cause Mortality (participants affected / at risk) | 22/129
Serious Adverse Events (participants affected / at risk) | 61/129
Other Adverse Events (participants affected / at risk) | 125/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belinostat (N=129)
Pneumonia (Infections and infestations) | 10
Pyrexia (General disorders) | 6
Infection (Infections and infestations) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Blood creatinine increased (Investigations) | 3
Multi-organ disorder (General disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Bronchitis (Infections and infestations) | 3
Cardiac failure (Cardiac disorders) | 2
Deep vein thrombosis (Vascular disorders) | 3
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Hypotension (Vascular disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Sepsis (Infections and infestations) | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Asthenia (General disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bronchitis bacterial (Infections and infestations) | 1
Central venous catheterisation (Surgical and medical procedures) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Device related infection (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Endocarditis (Infections and infestations) | 1
Euthanasia (General disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Gastrointestinal fungal infection (Infections and infestations) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Iliac artery occlusion (Vascular disorders) | 1
Impaired self-care (Psychiatric disorders) | 1
Liver function test abnormal (Investigations) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lung infection (Infections and infestations) | 1
Malaise (General disorders) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Pain (General disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pharyngitis (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Septic shock (Infections and infestations) | 1
Shock (Vascular disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Toxic cataract (Eye disorders) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Vasculitis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Chills (General disorders) | 1
Disease progression (General disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Bronchopneumopathy (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belinostat (N=129)
Nausea (Gastrointestinal disorders) | 55
Fatigue (General disorders) | 47
Pyrexia (General disorders) | 45
Anemia (Blood and lymphatic system disorders) | 41
Vomiting (Gastrointestinal disorders) | 37
Constipation (Gastrointestinal disorders) | 29
Diarrhea (Gastrointestinal disorders) | 28
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29
Edema Peripheral (General disorders) | 27
Rash (Skin and subcutaneous tissue disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Chills (General disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 21
Pruritus (Skin and subcutaneous tissue disorders) | 21
Blood Lactate Dehydrogenase Increased (Investigations) | 20
Decreased appetite (Metabolism and nutrition disorders) | 19
Headache (Nervous system disorders) | 19
Infusion Site Pain (General disorders) | 18
Hypokalemia (Metabolism and nutrition disorders) | 17
Abdominal Pain (Gastrointestinal disorders) | 14
Electrocardiogram QT Prolonged (Investigations) | 15
Hypotension (Vascular disorders) | 13
Phlebitis (Vascular disorders) | 12
Dizziness (Nervous system disorders) | 13
Asthenia (General disorders) | 12
Pain (General disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 13
Hyperglycemia (Metabolism and nutrition disorders) | 12
Bronchitis (Infections and infestations) | 9
Lymphopenia (Blood and lymphatic system disorders) | 11
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 11
Upper Respiratory Tract Infection (Infections and infestations) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Neuropathy Peripheral (Nervous system disorders) | 9
Aspartate Aminotransferase Increased (Investigations) | 11
Blood Creatinine Increased (Investigations) | 8
Platelet Count Decreased (Investigations) | 8
Flushing (Vascular disorders) | 9
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9
Insomnia (Psychiatric disorders) | 9
Alanine Aminotransferase Increased (Investigations) | 9
Hyperuricemia (Metabolism and nutrition disorders) | 8
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 8
Anxiety (Psychiatric disorders) | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 7
Nasopharyngitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 7
Blood Alkaline Phosphatase Increased (Investigations) | 7
Weight Decreased (Investigations) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No